CLINICAL TRIAL: NCT06720454
Title: Multiplex Immunofluorescence Staining of Pathological Tissue Microarray
Brief Title: Study on Single-cell Regulons Atlas of Pancreatic Ductal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Tiejun Ying (Other)
Responsible Party: Sponsor-Investigator, Tiejun Ying, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: YB M-05-01
Record Dates: First submitted 2024-12-01; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Molecular Prognostic Model; Regulons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The first purpose of this study is to reveal the gene regulatory network of pancreatic cancer by analyzing single-cell transcriptome sequencing data and to draw a pancreatic cancer regulator map. In addition, bulk transcriptome sequencing data are combined to construct and verify the genetic prognostic model of pancreatic cancer regulators, providing clinical tools for accurate prognostic stratification and personalized treatment of pancreatic cancer patients. The second purpose of this study is to explore the molecular mechanism by which the key oncogene in the gene prognostic model promotes pancreatic cancer advance. New ideas and scientific basis are provided for finding potential molecular targets for the treatment of pancreatic cancer. Thus, the investigators included a Tissue Microarray (TMA)-based cohort of 68 PDAC patient tissue samples. TMA was obtained from OUTDO BIOTECH (Shanghai, China). The study was approved by the institutional review board, and ethics document number is YB M-05-01.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic ductal adenocarcinoma
* With post-operative paraffin specimens

Exclusion Criteria:

* Other types of pancreatic cancer other than pancreatic ductal adenocarcinoma
* Without post-operative paraffin specimens or less than 20% of the paraffin sections contain cancerous tissue

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 68
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Intensity of immunofluorescence staining | From January 2019 to January 2024
  In this study, 68 pancreatic ductal adenocarcinoma tissues were used to detect the gene expression by multiple immunofluorescence staining

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China